CLINICAL TRIAL: NCT03528837
Title: Acute Kidney Injury in Neonates at NICU in Assiut University Children Hospital Descriptive Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Abdelrhman, Resident of neonatology, Assiut University
Other Study IDs: AKI neonates
Record Dates: First submitted 2018-04-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Neonatal Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosed as acute kidney injury: Sure diagnosed as acute kidney injury

SUMMARY:
Acute kidney injury (AKI) is a complex disorder with clinical manifestations ranging from mild dysfunction to complete anuric kidney failure. Its leads to sudden and rapid decline in renal excretory function within hours to days,accompanied by accumulation of nitrogenous waste products such creatinine,urea and other clinically un measured products

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an under-recognized morbidity of neonates; the incidence remains unclear due to the absence of a unified definition of AKI in this population and because previous studies have varied greatly in screening for AKI with serum creatinine and urine output assessments. Premature infants may be born with less than half of the nephrons compared with term neonates, predisposing them to chronic kidney disease (CKD) early on in life and as they age. AKI can also lead to CKD, and premature infants with AKI may be at very high risk for long-term kidney problems. AKI in neonates is often multifactorial and may result from prenatal, perinatal, or postnatal insults as well as any combination thereof.

ELIGIBILITY:
Inclusion Criteria:

* All cases of acute kidney injury in neonates who will be admitted to NICU Assiut University Children Hospital during the duration of the study.

Exclusion Criteria:

* Cases with chronic renal affection Any case with congenital anomalies

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study of cases of acute kidney injury in neonates and its causes and it's outcome
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosed as acute kidney injury | 10-21 days
  Diagnosis of acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university children hospital, Asyut, Egypt